CLINICAL TRIAL: NCT03248700
Title: Vitamin A Kinetics and Mathematical Modeling in American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-2008-0020; A074600 (Other: UW, Madison); AG&LSC/NUTRITIONAL SCI/NUTRITI (Other: UW, Madison)
Record Dates: First submitted 2017-08-08; First posted 2017-08-14 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Vitamin A Kinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin A tracer (Experimental): A stable isotope tracer of vitamin A was given orally.
  Interventions: Other: Vitamin A tracer

INTERVENTIONS:
Other: Vitamin A tracer — A stable isotope tracer of vitamin A was given orally.
  Other Names: 13C vitamin A; 13C retinyl acetate

SUMMARY:
Women were given a vitamin A tracer, and blood was sampled to determine individual and group vitamin A kinetics. Data were subsequently modeled using compartmental analysis to determine effects of study length on model outcomes.

DETAILED DESCRIPTION:
This is a longitudinal study in which American women were given an oral, stable isotope tracer of vitamin A, and blood was sampled in a staggered, serial design to determine individual and group vitamin A kinetics. Data were subsequently modeled using compartmental analysis, and study truncation analysis was performed on data to investigate the factor of study duration on resulting vitamin A kinetic models and outputs related to vitamin A metabolism.

ELIGIBILITY:
Inclusion Criteria:

* BMI (18.5 - 24.9 kg/m2)

Exclusion Criteria:

* Smoker
* Pregnant
* Trying to become pregnant
* Lactating
* Weight loss > 4.5 kg during the past 3 months.
* Actively trying to lose weight
* Inability to refrain from drinking alcohol when requested
* Amenorrhea
* Acute or chronic illness including hepatitis
* Current or previous history of anorexia or bulimia
* Concurrent participation in other studies
* Family member already enrolled in the study

Ages: 19 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2008-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Total traced vitamin A mass | Baseline through 152 days
  Total amount of endogenous vitamin A determined by mathematical model, (µmol).

SECONDARY OUTCOMES:
Compartmental model complexity | Baseline through 152 days
  Required number of compartments in mathematical model needed to adequately fit data.
Compartmental model fractional transfer coefficients | Baseline through 152 days
  Model parameters adjusted to fit analytical data. Represents the fractional transfer from one compartment to another in the model, (pools/d, represented as L(i,j), the fraction of compartment J transferred to compartment I per day).
Serum vitamin A half-life | Baseline through 152 days
  Half-life of vitamin A in serum, (d).
Vitamin A disposal rate | Baseline through 152 days
  Daily loss or utilization of vitamin A, (µmol/d).
Vitamin A equilibration time and partitioning | Baseline through 152 days
  Time taken for vitamin A to equilibrate with body stores, (d).
Vitamin A tracer partitioning | Baseline through 152 days
  Body partitioning of tracer between serum and extravascular compartment(s), relative to total tracee mass. Calculated as a ratio of tracer-to-tracee ratio (TTR) in serum and extravascular stores, (TTR serum / TTR stores).
Vitamin A dietary intake | Baseline
  Vitamin A dietary intake by food frequency questionnaire, (µg retinol activity equivalents/d).

CONTACTS AND LOCATIONS:
Overall Officials: Sherry A Tanumihardjo, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Department of Nutritional Sciences, University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gannon BM, Valentine AR, Davis CR, Howe JA, Tanumihardjo SA. Duration of Retinol Isotope Dilution Studies with Compartmental Modeling Affects Model Complexity, Kinetic Parameters, and Calculated Vitamin A Stores in US Women. J Nutr. 2018 Aug 1;148(8):1387-1396. doi: 10.1093/jn/nxy095. PMID 30137477